CLINICAL TRIAL: NCT05676528
Title: Kurzbewegungsintervention für Mitarbeitende Der Universität Bern
Brief Title: Exercise Intervention for Employees of the University of Bern
Acronym: WeMoveVirtual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-08-01; 2022-00970 (Other: Business Administration System for Ethics Committees (BASEC) number)
Record Dates: First submitted 2022-12-19; First posted 2023-01-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain; Musculoskeletal Diseases; Occupational Health; Efficiency; Exercise Therapy; Work Performance; Presenteeism
MeSH Terms: conditions — Neck Pain; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Exercise intervention
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — The participants will carry out a physiotherapeutic exercise intervention over a period of 6 weeks. The exercise intervention is stored in a smartphone app (PhysiApp) and consists of different neck and shoulder exercises. The investigators will provide the training material to the participants and they may keep it after the end of the study. Participants can choose which and how many exercises they would like to do. However, the investigators ask participants to exercise at least three times a week for 20 minutes each time (a total of one hour per week) and to document the training afterwards in the smartphone app. In the first, third and sixth week, the investigators train together with the participants via a virtual platform (e.g. video call via Microsoft Teams) so that the correct execution of the exercise can be checked and questions can be clarified.

SUMMARY:
As part of a Swiss National Science Foundation SNSF project (On-site multi-component intervention to improve productivity and reduce the economic and personal burden of neck pain in Swiss Office-Workers, NEXpro = Neck EXercises for productivity, SNSF no. 32003B_182389, BASEC no. 2019-01678), the investigators first developed a physiotherapeutic exercise intervention to improve the strength and mobility of the neck muscles. In the SNSF project NEXpro, the intervention took place on-site in the office. However, in view of the digital transformation, it is important to adapt the intervention delivery method to the new virtual work setting. The aims of the present project are therefore to implement, further develop and contextually adapt the exercise intervention in order to reduce musculoskeletal complaints and to reduce health-related presenteeism. The final product is a user-friendly virtual 6-week short exercise intervention that employees of the University of Bern can use independently, regardless of time and place. The effectiveness of the newly developed short exercise intervention (pain reduction, reduction of presenteeism) will be assessed during a short pilot phase.

ELIGIBILITY:
Inclusion Criteria:

* Employees of the Faculty of Human Sciences of the University of Bern who
* suffer from neck pain or would like to prevent neck pain
* are between 18 and 65 years of age
* understand German (written and oral)
* have a predominantly sedentary job
* have given written consent to participate in the study.

Note: Neither gender, age, education nor group affiliation play a role. The investigators particularly welcome participation from mid-level employees. If students are willing to participate, they may also do so, but this group will not be actively recruited.

Exclusion Criteria:

* Existing severe neck pain grade IV (neck trauma, neck injury, specific pathologies (e.g. congenital cervical anomalies, stenosis, radiculopathy), inflammatory conditions (e.g. rheumatoid arthritis), history of cervical surgery)
* If physical activity is contraindicated by the doctor for any reason (e.g. due to unresolved hypertension).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Work performance | 6 weeks
  Change in work performance from baseline. Work Productivity and Activity Impairment Questionnaire (i.e., work productivity loss). Min = 0, Max = 100. Higher score means worse (higher work productivity loss).

SECONDARY OUTCOMES:
Intensity of neck pain | Over the period of 6 weeks
  Change in neck pain from baseline. Numeric Rating Scale. Min = 0, Max = 10. Higher score means worse.
Intensity of back pain | Over the period of 6 weeks
  Change in back pain from baseline. Numeric Rating Scale. Min = 0, Max = 10. Higher score means worse.

OTHER OUTCOMES:
Level of physical activity | Over the period of 6 weeks
  Change of the level of physical activity from baseline. Questionnaire, single item (yes / no).
Sleep quality | Over the period of 6 weeks
  Change in sleep quality from baseline. Numeric Rating scale. Min = 1, Max = 5. Higher score means worse.
Work breaks | Over the period of 6 weeks
  Change in work breaks from baseline. Questionnaire, single item (number of work breaks)
General health status | Over the period of 6 weeks
  Change in general health status from baseline. Numeric Rating Scale. Min = 0, Max = 10. Higher score means better.
Mental health status | Over the period of 6 weeks
  Change in mental health status from baseline. Numeric Rating Scale. Min = 0, Max = 10. Higher score means better.
Flexibility | Over the period of 6 weeks
  Change in self-rated flexibility of the muscles from baseline. Numeric Rating Scale. Min = 0, Max = 10. Higher score means better.
Adherence to exercise 1 | Over the period of 6 weeks
  Number of exercise from baseline. Via PhysiApp. Higher score means higher number of exercise.
Adherence to exercise 2 | Over the period of 6 weeks
  Type of exercise from baseline. Via PhysiApp. Strengthening vs. non-strengthening.

CONTACTS AND LOCATIONS:
Overall Officials: Achim Elfering, Prof, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Faculty of Human Sciences, Institute of Psychology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No